CLINICAL TRIAL: NCT05098652
Title: Coaching Dementia Caregivers to Master Care-Resistant Behavior and Improve Coping Strategies
Brief Title: Coaching Dementia Caregivers to Master Care-Resistant Behavior
Acronym: CuRB-IT
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Alabama at Birmingham (Other)
Responsible Party: Principal Investigator, Rita A. Jablonski, Professor, University of Alabama at Birmingham
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: IRB-300007452
Record Dates: First submitted 2021-08-17; First posted 2021-10-28 (Actual); Last update posted 2025-04-25 (Actual); Status verified 2025-04

CONDITIONS: Care-resistant Behavior; Dementia
Keywords: dementia; care-resistant behavior; caregiver coping
MeSH Terms: conditions — Dementia

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Immediate Intervention (Experimental): Complete baseline survey, complete 3 weeks of daily diaries and intermittent survey, receive 12 weeks of CurB-IT, then complete 3 rounds of 21-day daily diaries and intermittent surveys while receiving attention during the 12-week intervals between daily diaries.
  Interventions: Behavioral: CuRB-IT
- Delayed intervention (Active Comparator): Complete baseline survey, complete 3 weeks of daily diaries, receive 12 weeks of attention, complete 3 weeks of daily diaries and 1 intermittent survey, receive 12 weeks of CurB-IT, then complete 2 rounds of 21-day daily diaries and intermittent surveys while receiving attention during the 12-week intervals between daily diaries.
  Interventions: Behavioral: CuRB-IT

INTERVENTIONS:
Behavioral: CuRB-IT — 9 1-hour coaching sessions delivered over a videoconferencing platform (Zoom); 6 delivered weekly, 3 delivered biweekly

SUMMARY:
266 family caregivers will be randomly assigned to either immediate intervention or delayed intervention groups. All caregivers will complete baseline surveys and 3 weeks of daily diaries. The immediate intervention group will receive 12 weeks of CuRB-IT. They will complete 3 rounds of 3-week daily diaries followed by an intermittent survey at 12 week intervals for the next 33 weeks. The delayed intervention group will receive 12 weeks of attention, complete 1 round of 3-week daily diaries followed by an intermittent survey, then complete 12 weeks of CuRB-IT, and complete 2 rounds of 3--week daily diaries followed by an intermittent survey at 12-week intervals for the next 18 weeks.

DETAILED DESCRIPTION:
The purposes of the delayed-intervention randomized clinical trial (N=266) are to:

Care-Resistant Behavior Internet Training (CuRB-IT).

1. examine the efficacy of CuRB-IT in increasing the self-efficacy of family caregivers of persons living with dementia to handle care-resistant behaviors (CRB);
2. further test the efficacy of CuRB-IT in improving caregivers coping strategies (a) among the experimental (immediate-intervention group) as compared to the control (delayed-intervention group) (between groups) and (b) within-person from pre- to post- intervention;
3. examine intervention decay at 3- and 6-months post intervention to determine performance of intervention and inform scheduling of booster sessions;
4. assess the efficacy of the CuRB-IT intervention in preventing onset of poor coping strategies by family caregivers;
5. test the hypothesized mechanism of action that increased CRB self-efficacy and use of CuRB-IT problem-focused coping strategies mediate the relationship between CRB stress appraisal and caregiving activities.

ELIGIBILITY:
Inclusion Criteria:

* 1)Caregiver of any race or gender who is aged >18 years
* 2) provides unpaid care,
* 3) cares for a spouse/common-law, sibling, parent or grandparent (or in-law, aged 60+ years),
* 4) lives with or shares cooking facilities with the care recipient,
* 5) Care recipient has mild cognitive impairment or dementia as identified using the Quick Dementia Rating System instrument,
* 6) the care provided consists of help with at least 2 Instrumental Activities of Daily Living or one Activity of Daily Living,
* 7) the care recipient is resistant to receiving assistance with, or refuses to do, at least one instrumental or activity of daily living

Exclusion Criteria:

* 1) persons who cannot speak/read English
* 2) who do not have reliable access to a smart phone or internet

Ages: 18 Years to 95 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 266 (Estimated)
Dates: Start 2023-04-01 (Actual); Primary Completion 2027-08-31 (Estimated); Study Completion 2027-09-30 (Estimated)

PRIMARY OUTCOMES:
Change in frequency of care-resistant behaviors and other dementia-related behaviors measured by a 19-item self-report scale (yes/no) for dementia family caregivers | Daily during weeks 1, 2, and 3
  Experimental and control
Change in frequency of care-resistant behaviors and other dementia-related behaviors measured by a 19-item self-report scale (yes/no) for dementia family caregivers | Daily during weeks 15, 16, and 17
  Experimental and control
Change in frequency of care-resistant behaviors and other dementia-related behaviors measured by a 19-item self-report scale (yes/no) for dementia family caregivers | Daily during weeks 37, 38, and 39
  Experimental and control
Change in frequency of care-resistant behaviors and other dementia-related behaviors measured by a 19-item self-report scale (yes/no) for dementia family caregivers | Daily during weeks 49, 50, and 51
  Experimental and control
Change in caregiver responses to dementia-related behaviors | Immediately after enrollment
  Experimental (immediate) and control (delayed intervention). Measured using yes/no responses to 8 items (2 from the Conflicts Tactics Scale Revised, 2 from the Conflicts Tactics Scale modified for Older Adults, and 4 from the Conflict Tactics Scale for Child Mistreatment).
Change in caregiver responses to dementia-related behaviors | Once at week 15
  Experimental (immediate) and control (delayed intervention). Measured using yes/no responses to 8 items (2 from the Conflicts Tactics Scale Revised, 2 from the Conflicts Tactics Scale modified for Older Adults, and 4 from the Conflict Tactics Scale for Child Mistreatment).
Change in caregiver responses to dementia-related behaviors | Once at week 37
  Experimental (immediate) and control (delayed intervention). Measured using yes/no responses to 8 items (2 from the Conflicts Tactics Scale Revised, 2 from the Conflicts Tactics Scale modified for Older Adults, and 4 from the Conflict Tactics Scale for Child Mistreatment).
Change in caregiver responses to dementia-related behaviors | Once at week 49
  Experimental (immediate) and control (delayed intervention). Measured using yes/no responses to 8 items (2 from the Conflicts Tactics Scale Revised, 2 from the Conflicts Tactics Scale modified for Older Adults, and 4 from the Conflict Tactics Scale for Child Mistreatment).
Change in caregiver self-efficacy coping skills | Immediately after enrollment
  Experimental (immediate) and control (delayed intervention). Measured using 14 items from the Brief Coping Scale.
Change in caregiver self-efficacy coping skills | Once at week 15
  Experimental (immediate) and control (delayed intervention). Measured using 14 items from the Brief Coping Scale.
Change in caregiver self-efficacy coping skills | Once at week 37
  Experimental (immediate) and control (delayed intervention). Measured using 14 items from the Brief Coping Scale.
Change in caregiver self-efficacy coping skills | Once at week 49
  Experimental (immediate) and control (delayed intervention). Measured using 14 items from the Brief Coping Scale.
Change in caregiver self-efficacy measured by selection of items from 10-item CurB-CuRB-IT Strategy checklist | Once at week 15
  Experimental (immediate)
Change in caregiver self-efficacy measured by selection of items from 10-item CurB-CuRB-IT Strategy checklist | Once at week 37
  Experimental (immediate)
Change in caregiver self-efficacy measured by selection of items from 10-item CurB-CuRB-IT Strategy checklist | Once at week 49
  Experimental (immediate)
Change in caregiver self-efficacy measured by selection of items from 10-item CurB-CuRB-IT Strategy checklist | Once at week 37
  Control (delayed)
Change in caregiver self-efficacy measured by selection of items from 10-item CurB-CuRB-IT Strategy checklist | Once at week 49
  Control (delayed)

CONTACTS AND LOCATIONS:
Overall Officials: Rita A Jablonski, PhD, Principal Investigator — University of Alabama at Birmingham
Locations (1):
- University of Alabama at Birmingham, Birmingham, Alabama, United States

IPD SHARING:
Plan to Share IPD: Yes
All research data produced by this project will be self-archived at the University of Michigan's NIA-funded National Archive of Computerized Data on Aging. The storage of our research product here will permit many researchers free access to our data in perpetuity. Our archived study will principally include our original (but anonymized) databases as well as any "cleaned," computed, and recoded measures that we produce for or is produced by our analysis. Our project deliverables will include the quantitative databases, a well-documented statistical packaging (SPSS) system file with variable and values labels, a data user guide that includes all SPSS and related computational and analysis syntax code, summary statistics (frequency distributions, means, etc.) for all quantitative variables, a copy of applicable subject consent form, human subject application and the institutional review board (IRB) approval letter, and a blank copy of the survey instrument and interviewer guide.
Supporting Information: Study Protocol, SAP, ICF, Analytic Code
Time Frame: 6 months after conclusion of study; in perpetuity
Access Criteria: 1) a commitment only to use the data for research purposes and not to identify any individual participant; 2) a commitment to securing the data using appropriate computer technology; and 3) a commitment to destroy or return the data after analyses are completed.